CLINICAL TRIAL: NCT04404127
Title: Standard Induction With Basiliximab Versus No-Induction in Low Immunological Risk Kidney Transplant Recipients - Prospective Randomized Double Blind Controlled Clinical Trial
Brief Title: Standard Induction With Basiliximab Versus No-Induction in Low Immunological Risk Kidney Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Aziza Ajlan, Aziza A. Ajlan, B.Sc. Pharm. BCPS. Clinical pharmacy specialist- Solid Organ Transplant, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAC # 2191177
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Kidney Transplantation
Keywords: basiliximab; Rejection; De no vo donor specific antibodies; Low immunological risk; Induction
MeSH Terms: conditions — Rejection, Psychology | interventions — Basiliximab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The trial will be blinded with respect to Basiliximab induction allocation. The study will be blinded to subjects and site study investigators, with the following exceptions:
  A single pharmacist A single biostatistician Patients with receive either basiliximab or an intravenous piggyback (IVPB) with normal saline depending on their allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No induction Arm (Placebo Comparator)
  Interventions: Other: Normal Saline
- Induction with basiliximab (Active Comparator)
  Interventions: Drug: Basiliximab 20 milligram [Simulect]

INTERVENTIONS:
Drug: Basiliximab 20 milligram [Simulect] — Basiliximab
  Arms: Induction with basiliximab
Other: Normal Saline — No-Induction
  Arms: No induction Arm

SUMMARY:
Background:

Induction therapy with IL-2 receptor antagonist (IL2-RA) is recommended as a first line agent in low immunological risk kidney transplant recipients. However, the role of IL2-RA in the setting of tacrolimus-based immunosuppression has not fully investigated

Aims:

To compare different induction therapeutic strategies with 2 doses of Basiliximab vs. no induction) in low immunologic risk kidney transplant recipients as per KFSHRC protocol (Appendix 2)

Methods:

Prospective, randomized, double blind, non-inferiority, controlled clinical trial

Expected Outcomes:

1. Primary outcomes:

   Biopsy proven acute rejection within first year following transplant
2. Secondary outcomes:

   1. Patient and graft survival at 1 year
   2. Estimated glomerular filtration rate (eGFR) at 6 months and at 12 months
   3. Emergence of de novo donor specific antibodies (DSAs)

ELIGIBILITY:
Inclusion Criteria:

* • Male or female ≥ 18 years

  * Living donor
  * Low immunological risk (defined as):

    1. First (primary) transplant
    2. ≤ 4 antigen mismatches (HLA matching scheme)
    3. Negative HLA Ab screening

Exclusion Criteria:

* • High immunological risk

  * HLA identical or zero mismatched transplants
  * Receiving cyclosporin as primary maintenance immunosuppressant
  * Human immunodeficiency virus (HIV) co-infection
  * Pregnant or nursing female
  * Has received an investigational medication within the past 30 days
  * Has a known contraindication to the administration of Basiliximab
  * Suspected or known to have a serious infection
  * Multi-organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Rate of biopsy proven acute rejection within first year following transplant | 1 year after transplant

SECONDARY OUTCOMES:
Rate of graft survival at 1 year | 1 year after transplant
Rate of decline in eGFR at 6 months and at 12 months | 1 year after transplant
Rate of emergence of de novo donor specific antibodies (DSAs) | 1 year after transplant

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research Centre (KFSHRC), Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No